CLINICAL TRIAL: NCT04816500
Title: Study of Efficacy and Safety of Remote Ischemic Conditioning on Cerebral Small Vessel Disease
Brief Title: Remote Ischemic Conditioning on Cerebral Small Vessel Disease
Acronym: RIC-SVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Study of Efficacy and Safety of remote ischemic conditioning on cerebral small vessel disease, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Capital Medical U
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Cerebral Small Vessel Diseases; Remote Ischemic Conditioning
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIC group (Experimental): Device: Remote ischemic conditioning RIC is a non-invasive therapy that performed by an electric autocontrol device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on one arm. The procedure will be performed twice daily for consecutive 1 year after enrollment.
  Interventions: Device: Automatic ischemic conditioning treatment instrument
- Regular treatment (Other)
  Interventions: Drug: Regular treatment

INTERVENTIONS:
Device: Automatic ischemic conditioning treatment instrument — RIC is a non-invasive therapy that performed by an electric autocontrol device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on one arm. The procedure will be performed twice daily for consecutive 1 year after enrollment.
  Arms: RIC group
Drug: Regular treatment — Antiplatelet agents and statins administration, vascular risk factors control.
  Arms: Regular treatment

SUMMARY:
This trial is a randomized, controlled, single-center, double-blind trial. Cerebral small vessel disease (CSVD) patients will be recruited and randomized into RIC or control group.The protective effect of remote ischemic conditioning (RIC) on CSVD will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. 45-80 years old, and gender not limited;
2. patient and/or caregiver report of cognitive declines with regard to memory and/or other cognitive domains lasting for at least 3 months;
3. neither normal nor demented on the basis of the criteria of the Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) with normal or slightly impaired activities of daily living9, with Mini-mental State Examination (MMSE) score ≥ 20 (primary school) or ≥ 24 (junior school or above)10 and Montreal Cognitive Assessment (MoCA) score ≤ 26;
4. the presence of lacunes and/or WMHs and/or CMBs on MRI
5. absence of vascular narrowing >50% luminal diameter that could cause hemodynamic changes (MFV>90 cm/s for the intracranial internal carotid artery, 100 cm/s for MCA, >80 cm/s for basilar artery [BA] or vertebral artery) measured by TCD

Exclusion Criteria:

1. clinical manifestations indicating that the patient was at the end-stage of cSVD;
2. hereditary or inflammatory small vessel disorders
3. cerebral venous injury or changes;
4. diagnosis of nervous system degenerative diseases Alzheimer's disease, DLB, frontotemporal dementia (FTD), and so on;
5. history of intracranial hemorrhage or significant bleeding in other parts of the body
6. brain tumor, psychoses, or acute stroke within 6 months;
7. cardiogenic embolism;
8. significant bleeding coagulation dysfunction;
9. serious liver and kidney function is not complete, malignant tumor, or serious diseases need to medical intervention or surgery;
10. any soft tissue or vascular injury, and any disease of the extremities that may contraindicate RIC;
11. pregnant women;
12. life expectancy<6 months;
13. refused to sign a consent form, poor compliance, or not to cooperate to complete whole treatment, and so on.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of volume of WMHs | From baseline to 1 year treatment
  The volume of WMHs was measured on Flairs and DTI. By calculating the mean diffusivity (MD) and FA of water diffusion, DTI can assess the integrity and connectivity of WM tissue from a network perspective, and reconstruct the distribution of WM pathways in the brain three-dimensionally.

SECONDARY OUTCOMES:
Changes in hemodynamic parameters on TCD. | From baseline to 1 year treatment
  The peak systolic, mean, and end diastolic blood flow velocities (BFV) at the most proximal segment of bilateral MCAs, BA were measured by TCD
Changes of cognition evaluation on MoCA. | From baseline to 1 year treatment
  The Beijing version of MoCA were used to evaluate to evaluate the cognitive functions of patients, referring to the degree of an individual's capacity with respect to orientation, memory, calculation, language, execution and visuospatial function and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu hospital;Capital Medical University, Beijin, China

IPD SHARING:
Plan to Share IPD: Undecided